CLINICAL TRIAL: NCT03430752
Title: Comparing the Impact of Cancer and Treatment-related Effects on the Psychological Well-Being and Quality of Life Between Survivors of Childhood Solid Tumors and Leukemia
Brief Title: Comparing the Impact of Cancer on Quality of Life Between Survivors of Childhood Solid Tumors and Leukemia
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW 17-331 (2)
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Childhood Solid Tumor
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivors of Childhood Solid Tumors: Survivors of Childhood Solid Tumors were invited to fill in a set of questionnaires.
  Interventions: Other: questionnaires
- Survivors of Childhood Leukemia: Survivors of Childhood Leukemia were invited to fill in a set of questionnaires.
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — Participants were asked to respond to the questionnaires including the Chinese version of the Paediatric Quality of Life Inventory 4.0 Generic Core Scale (PedsQL 4.0), the Chinese version of the Center for Epidemiological Studies Depression Scale for Children (CES-DC), the Chinese version of Rosenberg self-esteem scale, the Chinese version of the Herth Hope Index (HHI) and the Chinese version of Resilience Scale for Children (RS10).

SUMMARY:
The aim of the study is to examine the impact of cancer and treatment-related effects on the physical and psychosocial well-being and quality of life among Hong Kong Chinese survivors of childhood solid tumors.

DETAILED DESCRIPTION:
In general, cancer can be divided into two main categories: blood cancer and solid tumors. Leukemia refer to the cancers in blood while solid tumors refer to the cancers which involve the formation of an abnormal mass without any liquid or cysts. Patients suffer from leukemia are usually have better prognosis which result in better psychological well-being when compared with those suffer from solid tumors (Rodin et al., 2010). The development of solid tumors in children is different from that in adult. Some of the solid tumors such as osteosarcoma, neuroblastoma, rhabdomyosarcoma, Wilms' tumor and retinoblastoma are exclusively found in children. Other types of solid tumors such as brain tumor can also be found in children.

Yet, most of recent studies in Hong Kong have focused in general childhood cancer survivors or their family members but no study has been conducted to focus on the physical and psychological well-being of survivors of childhood solid tumors (Li, Lopez, Chung, Ho, & Chiu, 2013; Wills, 2009). Therefore, the quality of life and psychological well-being of solid tumors survivors are always be overestimated. The actual psychological needs of solid tumors survivors may be overlooked. There is thus an imperative need to investigate the impact of cancer and treatment-related effects on the physical and psychosocial well-being and quality of life among Hong Kong Chinese survivors of childhood solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* (1) Hong Kong Chinese under the age of 30 years at the time of study participation;
* (2) diagnosed with solid tumors or hematological malignancies under the age of 19 years;
* (3) completed the entire course of treatment for at least 6 months;
* (4) able to speak fluent Cantonese and read Chinese.

Exclusion Criteria:

* Survivors with secondary malignancy, organic cause psychosis, cognitive or learning problems, or under active cancer treatment will be excluded from this study.

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Hong Kong Chinese under the age of 19 years who completed the entire course of treatment at least 6 months and were diagnosed with childhood solid tumors or leukemia under the age of 19 years.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Quality of Life at baseline | Baseline
  The Pediatric Quality-of-Life Inventory 4.0 Generic core sales (PedsQL 4.0) consists of 23 items which are designed to measure the quality of life in four particular domains including physical ability, psychological states, social relationships and school functioning. PedsQL 4.0 is a five-point Likert scale for patients to response regarding to the experience over the last month. Higher scores represent better quality of life. Participants will be asked to respond to the Pediatric Quality-of-Life Inventory 4.0 Generic core sales (PedsQL 4.0) at baseline.

SECONDARY OUTCOMES:
Levels of self-esteem at baseline | Baseline
  The self-esteem of the participants will be measured by the Chinese version of the Rosenberg Self-esteem Scale (RSES). RSES consists of 10 items with a four-point response Likert scale ranging from 1 (strongly agree) to 4 (strongly disagree) and the total scores is ranging from 10 to 40. Higher scores represent higher levels of self-esteem. Participants will be asked to respond to the Chinese version of the Rosenberg Self-esteem Scale (RSES) at baseline.
Number of depressive symptoms at baseline | Baseline
  The number of depressive symptoms of the participants will be measured by the Center for Epidemiological Studies - Depression Scale for children (CES-DC). It is able to assess the numbers of depressive symptoms due to the experience of past week. The scale consists of 20 items with four-point Likert scale for patients to response and the total score is ranging from 0 to 60. Higher scores represent greater numbers of depressive symptoms while lower scores represent fewer numbers of depressive symptoms. Participants will be asked to respond to the Center for Epidemiological Studies - Depression Scale for children (CES-DC) at baseline.
Level of sense of hope at baseline | Baseline
  The sense of hope of the participants will be measured by the Chinese version of Herth Hope Index (HHI). It is a 12-item psychometric scale to measure the sense of hope. Each item contains four-point scale ("strong disagree" = "1", "disagree" = "2", "agree" = "3", "strong agree" = "4"). The total score of the 12 items ranging from 12 to 48 and higher scores imply increasing hopefulness. Participants will be asked to respond to the Chinese version of the Herth Hope Index (HHI) at baseline.
Resilience ability at baseline | Baseline
  Resilience Scale for Children (RS10) is a 10-item scale to assess the adjustment ability for adapting adverse conditions such as cancer. The scale consists of 10 items with four-point Likert scale ("not at all like me"= "1", "not much like me" = "2", "somewhat like me" = "3", "a lot like me" = "4"). The total score is ranging from 10 to 40 which higher scores represent higher level of resilience. Participants will be asked to respond to the Chinese version of the Resilience Scale for Children (RS10) at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No